CLINICAL TRIAL: NCT06897306
Title: Surgery Significantly Improves the Prognosis of Locally Advanced Gastric-type Endocervical Adenocarcinoma: a Population-based Cohort Study
Brief Title: Gastric-type Endocervical Adenocarcinoma: a Population-based Cohort Study
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2025-057-01
Record Dates: First submitted 2025-02-06; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Uterine Cervical Neoplasms; Surgery; Therapy; Locally Advanced Cervical Carcinoma
Keywords: Uterine Cervical Neoplasms; cervical cancer; Gastric - type Mucinous Adenocarcinoma; surgery
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery — The patient underwent surgery.

SUMMARY:
This study aims to collect data of patients with Gastric-type Endocervical Adenocarcinoma from the SEER database, analyze the related prognostic factors and treatment patterns of Gastric-type Endocervical Adenocarcinoma, and explore the impact of surgical treatment on the prognosis of locally advanced Gastric-type Endocervical Adenocarcinoma.

DETAILED DESCRIPTION:
This study aims to collect data of patients with Gastric - type Endocervical Adenocarcinoma from the SEER database, analyze the related prognostic factors and treatment patterns of patients with Gastric - type Endocervical Adenocarcinoma, and explore the impact of surgical treatment on the prognosis of locally advanced Gastric - type Endocervical Adenocarcinoma.

Study subjects: Patients diagnosed with Gastric - type Endocervical Adenocarcinoma were identified using the SEER database and SEER*Stat 8.4.2 software. The search scope was the "SEER Research Plus Data, 17 Registries, Nov 2021 sub (2000 - 2019)" database, and the screening criteria included "Site and Morphology, Analytic Behavior Recode = Malignant" and "Site and Morphology, ICD - O - 3 / WHO 2008 Recode Site = Cervix". Patients with cervical Gastric - type Endocervical Adenocarcinoma were selected from the database.

Outcome measures: Overall survival (OS): The time from diagnosis to death of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Gastric - type Endocervical Adenocarcinoma were identified using the SEER database and SEER*Stat 8.4.2 software. The search scope was the "SEER Research Plus Data, 17 Registries, Nov 2021 sub (2000 - 2019)" database. The screening criteria included "Site and Morphology, Analytic Behavior Recode = Malignant" and "Site and Morphology, ICD - O - 3 / WHO 2008 Recode Site = Cervix". Patients with Gastric - type Endocervical Adenocarcinoma in the database were selected.

Exclusion Criteria:

* Patients with a survival time of 0 or unknown.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Surveillance, Epidemiology, and End Results (SEER) database is a comprehensive source of population - based cancer incidence and survival data in the United States. The population covered by the SEER database is diverse and representative of the broader U.S. population. It includes individuals from various racial and ethnic backgrounds, age groups, and geographic regions. The data are collected from 17 population - based cancer registries, which cover approximately 28% of the U.S. population. This allows for the analysis of cancer - related outcomes and trends across different demographic and socioeconomic groups, providing valuable insights into the burden of cancer and the effectiveness of cancer - related interventions in a population - based setting.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | The time from diagnosis to death of the patient，Assessed up to 227 months
  The time from diagnosis to death of the patient.

SECONDARY OUTCOMES:
Vital status recode(study cutoff used) | up to 227 months
  Any patient that dies after the follow-up cut-off date is recoded to alive as of the cut-off date.

CONTACTS AND LOCATIONS:
Overall Officials: Huaiwu Lu, Study Director — The Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- The Sun Yat-Sen Memorial Hospital of Sun Yat-Sen Universit, Guangzhou, Guangdong, China